CLINICAL TRIAL: NCT04225988
Title: A Prospective, Pilot Trial to Compare the Efficacy of Tacrolimus Extended-Release (Envarsus XR) to Tacrolimus Immediate-Release on Suppression of Donor-Specific Antibodies in HLA Sensitized Kidney Transplant Recipients
Brief Title: Comparison of Tacrolimus Extended-Release (Envarsus XR) to Tacrolimus Immediate-Release in Human Leukocyte Antigen (HLA) Sensitized Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Veloxis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Edmund Huang, Staff Physician II, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00054474
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-06

CONDITIONS: Kidney Transplant Rejection
Keywords: kidney transplant; rejection; donor-specific antibodies
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Extended-release tacrolimus (Experimental): Kidney transplant recipients will receive extended-release tacrolimus in addition to standard-dose mycophenolate and prednisone for maintenance immunosuppression.
  Interventions: Drug: Extended-release tacrolimus
- Immediate-release tacrolimus (Active Comparator): Kidney transplant recipients will receive immediate-release tacrolimus in addition to standard-dose mycophenolate and prednisone for maintenance immunosuppression.
  Interventions: Drug: Immediate-release tacrolimus

INTERVENTIONS:
Drug: Extended-release tacrolimus — Patients will receive the extended-release formulation of tacrolimus for maintenance immunosuppression.
  Arms: Extended-release tacrolimus
Drug: Immediate-release tacrolimus — Patients will receive the immediate-release formulation of tacrolimus for maintenance immunosuppression.
  Arms: Immediate-release tacrolimus

SUMMARY:
This is a randomized, open-label, controlled clinical trial designed to compare clinical outcomes after kidney transplantation using extended-release tacrolimus (Envarsus XR) versus immediate tacrolimus among highly-sensitized kidney transplant recipients. Outcomes to be assessed include the incidence of biopsy-proven acute rejection at 12 months, the presence of de novo and pre-existing donor-specific HLA antibodies, estimated glomerular filtration rate, and the level of donor-derived cell-free DNA.

DETAILED DESCRIPTION:
Extended-release tacrolimus (Envarsus XR) received FDA approval in July, 2015 for the prevention of allograft rejection in kidney transplantation on the basis of two separate phase 3 trials of de novo and stable kidney transplant recipients that demonstrated non-inferiority to immediate-release tacrolimus for the composite outcome of death, graft failure, biopsy-proven acute rejection, or loss to follow-up within 12 months (1,2).

Both phase 3 trials involved mostly low immunologic risk recipients with follow-up to one year. It has been previously shown that the incidence of de novo donor-specific antibodies (DSA) in the first year after kidney transplant in low-immunologic patients is low, developing in only 2%-11% of unsensitized de novo kidney transplant recipients (3-6). Donor-specific antibodies (DSA) are the primary mediator of antibody-mediated rejection and their development after transplant is a major risk factor for late allograft failure (7). It is now believed that antibody-mediated rejection is the most common cause of late allograft failure (8,9). However, neither of the two phase 3 trials were able to adequately assess the effect of Envarsus XR on the development of donor specific antibodies and therefore, the efficacy of Envarsus XR in higher immunologic risk recipients is not known. Therefore, a comparative study of extended- and immediate-release tacrolimus in highly-sensitized recipients is warranted.

This is a randomized, open-label, controlled clinical trial designed to compare clinical outcomes after kidney transplantation using extended-release tacrolimus (Envarsus XR) versus immediate tacrolimus among highly-sensitized kidney transplant recipients. Twenty patients will be enrolled, with ten assigned to each study arm. Outcomes to be assessed include the incidence of biopsy-proven acute rejection at 12 months, the presence of de novo and pre-existing donor-specific HLA antibodies, estimated glomerular filtration rate, and the level of donor-derived cell-free DNA.

ELIGIBILITY:
Inclusion Criteria:

1. Recipient of a deceased or living donor kidney allograft
2. Patients must have undergone desensitization with Intravenous Immunoglobulin (IVIG) and rituximab with or without plasma exchange prior to transplant or be administered IVIG and rituximab peri-operatively (within seven days of transplant) post-transplant
3. Age 18 and over
4. Able to understand and provide informed consent
5. At transplant, patient must have an acceptable crossmatch [as defined by a T- or B-flow crossmatch ≤ 225 median channel shift (MCS)] from a non-HLA identical donor. A negative crossmatch is defined as a T pronase flow crossmatch < 70 MCS or a T- flow crossmatch < 50 MCS and a B pronase flow crossmatch <130 MCS or a B-flow crossmatch <100 MCS.

Exclusion Criteria:

1. Recipients of a dual simultaneous kidney/liver, kidney/heart, kidney/lung, or kidney/pancreas transplant.
2. History of hypersensitivity to any of the study drug or to drugs of similar chemical classes.
3. Patients with a clinically significant systemic infection within 30 days prior to transplant.
4. Patients who have any history of a surgical or medical condition that may affect absorption of drug, such as severe diarrhea, active peptic ulcer disease, or uncontrolled diabetes mellitus, which in the opinion of the investigator at the time of enrollment, might significantly alter the absorption, distribution, metabolism and/or excretion of study medication.
5. Women of childbearing potential who are either pregnant, lactating, planning to become pregnant during this trial, or with a positive serum or urine pregnancy test. Women of childbearing potential must be willing to agree to contraceptive practices.
6. Patients who are Polymerase Chain Reaction (PCR) positive for hepatitis B, hepatitis C, or HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data with other researchers.

REFERENCES:
- [Background] Budde K, Bunnapradist S, Grinyo JM, Ciechanowski K, Denny JE, Silva HT, Rostaing L; Envarsus study group. Novel once-daily extended-release tacrolimus (LCPT) versus twice-daily tacrolimus in de novo kidney transplants: one-year results of Phase III, double-blind, randomized trial. Am J Transplant. 2014 Dec;14(12):2796-806. doi: 10.1111/ajt.12955. Epub 2014 Oct 2. PMID 25278376
- [Background] Bunnapradist S, Ciechanowski K, West-Thielke P, Mulgaonkar S, Rostaing L, Vasudev B, Budde K; MELT investigators. Conversion from twice-daily tacrolimus to once-daily extended release tacrolimus (LCPT): the phase III randomized MELT trial. Am J Transplant. 2013 Mar;13(3):760-9. doi: 10.1111/ajt.12035. Epub 2012 Dec 21. PMID 23279614
- [Background] Everly MJ, Rebellato LM, Haisch CE, Ozawa M, Parker K, Briley KP, Catrou PG, Bolin P, Kendrick WT, Kendrick SA, Harland RC, Terasaki PI. Incidence and impact of de novo donor-specific alloantibody in primary renal allografts. Transplantation. 2013 Feb 15;95(3):410-7. doi: 10.1097/TP.0b013e31827d62e3. PMID 23380861
- [Background] Hidalgo LG, Campbell PM, Sis B, Einecke G, Mengel M, Chang J, Sellares J, Reeve J, Halloran PF. De novo donor-specific antibody at the time of kidney transplant biopsy associates with microvascular pathology and late graft failure. Am J Transplant. 2009 Nov;9(11):2532-41. doi: 10.1111/j.1600-6143.2009.02800.x. PMID 19843031
- [Background] Schinstock CA, Cosio F, Cheungpasitporn W, Dadhania DM, Everly MJ, Samaniego-Picota MD, Cornell L, Stegall MD. The Value of Protocol Biopsies to Identify Patients With De Novo Donor-Specific Antibody at High Risk for Allograft Loss. Am J Transplant. 2017 Jun;17(6):1574-1584. doi: 10.1111/ajt.14161. Epub 2017 Jan 25. PMID 27977905
- [Background] Wiebe C, Gibson IW, Blydt-Hansen TD, Pochinco D, Birk PE, Ho J, Karpinski M, Goldberg A, Storsley L, Rush DN, Nickerson PW. Rates and determinants of progression to graft failure in kidney allograft recipients with de novo donor-specific antibody. Am J Transplant. 2015 Nov;15(11):2921-30. doi: 10.1111/ajt.13347. Epub 2015 Jun 10. PMID 26096305
- [Background] Loupy A, Hill GS, Jordan SC. The impact of donor-specific anti-HLA antibodies on late kidney allograft failure. Nat Rev Nephrol. 2012 Apr 17;8(6):348-57. doi: 10.1038/nrneph.2012.81. PMID 22508180
- [Background] Sellares J, de Freitas DG, Mengel M, Reeve J, Einecke G, Sis B, Hidalgo LG, Famulski K, Matas A, Halloran PF. Understanding the causes of kidney transplant failure: the dominant role of antibody-mediated rejection and nonadherence. Am J Transplant. 2012 Feb;12(2):388-99. doi: 10.1111/j.1600-6143.2011.03840.x. Epub 2011 Nov 14. PMID 22081892
- [Background] Einecke G, Sis B, Reeve J, Mengel M, Campbell PM, Hidalgo LG, Kaplan B, Halloran PF. Antibody-mediated microcirculation injury is the major cause of late kidney transplant failure. Am J Transplant. 2009 Nov;9(11):2520-31. doi: 10.1111/j.1600-6143.2009.02799.x. PMID 19843030

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female HLA sensitized (HS) renal transplantation patients, 18 years of age and over, receiving a deceased or living donor kidney allograft may enter the study. Twenty patients will be enrolled at Cedars-Sinai Medical Center (CSMC) for this pilot study. Patients who discontinue the study prematurely will not be replaced.
Pre-assignment Details: Of the total 28 participants ages 18 and older screened, 20 were enrolled in this single-center, open-label, randomized controlled trial design pilot study.
Period: Overall Study
Arm/Group | Extended-release Tacrolimus | Immediate-release Tacrolimus
Started | 10 | 10
Completed | 8 | 10
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Extended-release Tacrolimus | Immediate-release Tacrolimus | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (15.0200) | 46.1 (11.6376) | 47.85 (13.2000)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 3 | 6 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 6 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 7 | 10 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Biopsy-proven Acute Rejection
Description: To assess whether the occurence of biopsy-proven acute rejection within 12 months of transplant is comparable between HS patients maintained on Envarsus XR and immediate-release tacrolimus.
Time Frame: 12 months
Population: All participants who completed their 12 month visit were assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-release Tacrolimus | Immediate-release Tacrolimus
Number analyzed (Participants) | 8 | 10
Participants | 1 | 2

2. Secondary Outcome: Number of Participants With de Novo Donor-specific Antibodies
Description: To assess the number of participants who developed a presence of de novo donor-specific antibodies developing between Envarsus XR-treated and immediate-release tacrolimus-treated HS recipients.
Time Frame: 12 months
Population: All participants who completed their 12 month visit were assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-release Tacrolimus | Immediate-release Tacrolimus
Number analyzed (Participants) | 8 | 10
Participants | 1 | 1

3. Secondary Outcome: Number of Persistent Pre-existing Donor-specific Antibodies
Description: To assess the number of participants who had persistent pre-existing donor-specific antibodies at 12 months in the Envarsus XR-treated and immediate-release tacrolimus-treated groups.
Time Frame: 12 months
Population: All participants who completed their 12 month visit were assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-release Tacrolimus | Immediate-release Tacrolimus
Number analyzed (Participants) | 8 | 10
Participants | 1 | 2

4. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR; Chronic Kidney Disease (CKD)-Epi Equation)
Description: To assess the mean eGFR (using the CKD-Epi equation) between Envarsus XR-treated and immediate-release tacrolimus-treated HS recipients.
Time Frame: 12 months
Population: All participants who completed their 12 month visit were assessed.
Measure: Median (Inter-Quartile Range); unit: ml/min/1.73 m2
Arm/Group | Extended-release Tacrolimus | Immediate-release Tacrolimus
Number analyzed (Participants) | 8 | 10
ml/min/1.73 m2 | 58 [50 to 74] | 59 [38 to 67]

5. Secondary Outcome: Level of Donor-derived Cell-free DNA (Allosure)
Description: To assess the mean percentage of donor-derived cell-free DNA (Allosure) between Envarsus XR-treated and immediate-release tacrolimus-treated HS recipients.
Time Frame: 6 months and 12 months
Population: All participants who completed their 12 month visit were assessed.
Measure: Mean (Standard Deviation); unit: % donor-derived cell-free DNA
Arm/Group | Extended-release Tacrolimus | Immediate-release Tacrolimus
Number analyzed (Participants) | 8 | 10
% donor-derived cell-free DNA
  6 Months | 0.599 (0.688) | 1.343 (1.180)
  12 Months | 1.166 (0.926) | 2.093 (1.681)

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse events and severe adverse events were collected and reported in all enrolled participants who received extended-release or immediate-release Tacrolimus.
Arm/Group | Extended-release Tacrolimus | Immediate-release Tacrolimus
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 6/10 | 6/10
Other Adverse Events (participants affected / at risk) | 4/10 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended-release Tacrolimus (N=10) | Immediate-release Tacrolimus (N=10)
Vaginal abscess (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Transplant pyelonephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fever (Infections and infestations) | 2 (2) | 0 (0)
Thoracic back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (2) | 0 (0)
Acute hemorrhage (Infections and infestations) | 0 (0) | 1 (1)
Enterococcus bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0)
Post transplantation diabetes melitus (PTDM) (Endocrine disorders) | 1 (1) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urinary tract infection (UTI) (Infections and infestations) | 2 (4) | 0 (0)
Nausea and Vomiting (General disorders) | 1 (1) | 0 (0)
Diarrhea (General disorders) | 1 (1) | 0 (0)
Elevated serum creatinine (Renal and urinary disorders) | 1 (2) | 1 (1)
Secondary acute idney injury (AKI) (Renal and urinary disorders) | 1 (2) | 0 (0)
Hypogamma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dehydration (General disorders) | 1 (1) | 0 (0)
Abnormal labs (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended-release Tacrolimus (N=10) | Immediate-release Tacrolimus (N=10)
Nausea (General disorders) | 0 (0) | 1 (1)
Dehydration (General disorders) | 0 (0) | 1 (1)
Right lower quardrant abdominal pain (General disorders) | 0 (0) | 1 (1)
Vomitting (General disorders) | 0 (0) | 1 (1)
Elevated serum creatinine (Renal and urinary disorders) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypotension (General disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3)
BK Viremia (Infections and infestations) | 1 (1) | 0 (0)
Antibody-mediated rejection (Renal and urinary disorders) | 0 (0) | 1 (1)
Wrist abscess (Infections and infestations) | 0 (0) | 1 (1)
Norcadia nova (Infections and infestations) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hair loss (General disorders) | 1 (1) | 0 (0)
Cough (Infections and infestations) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Loose stools (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Increased Allosure (Renal and urinary disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size; Early withdrawal of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-03): https://cdn.clinicaltrials.gov/large-docs/88/NCT04225988/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-17): https://cdn.clinicaltrials.gov/large-docs/88/NCT04225988/ICF_001.pdf